CLINICAL TRIAL: NCT01119170
Title: Safety Assessment of a Starter Formula Containing D-lactate Producing Probiotics
Brief Title: Safety of D-lactate Producing Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.51.INF
Record Dates: First submitted 2010-04-27; First posted 2010-05-07 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Acidosis
Keywords: nutrition; infant formula; probiotics
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control starter formula (Placebo Comparator)
  Interventions: Other: Starter formula
- D-lactate probiotics (Experimental)
  Interventions: Other: starter formula with D-lactate producing probiotics

INTERVENTIONS:
Other: Starter formula — standard starter formula given from birth to 6 months of age
  Arms: control starter formula
Other: starter formula with D-lactate producing probiotics — starter formula containing probiotics given from birth to 6 months of age
  Arms: D-lactate probiotics

SUMMARY:
In this study the investigators want to test the safety of D-lactate producing probiotics in babies from birth to 1 month of age. Previous data demonstrated no increase in urinary D-lactate in 4 month old infants supplemented with D-lactate producing probiotics. The primary purpose of this study is to evaluate the influence of D-lactate producing probiotics on D-lactate excretion in young infants during the neonatal period (days 0 - 28).

DETAILED DESCRIPTION:
Lactate, in addition to being found in more common fermented foods of today, such as yogurt, lactate, in its two stereoisomer forms, known as the D (dextrorotary) or L (levorotary) is also produced in the colon through the normal fermentative process of lactic acid producing bacteria. Both D-lactate and L-lactate produced by these microbes are metabolized by enzymes within human cells and do not typically pose an acid-base risk by reducing pH to a threatening degree in healthy individuals.

However, the specific dehydrogenase that converts D-lactate to pyruvate is far less active than that for L-lactate, and it has been suggested that very young infants may be a vulnerable group for D-lactic acidosis. Previous data have shown that urinary D-/L- lactate excretion were not significantly different between 2 groups of 4 month old infants taking a control formula or a formula containing D-lactate producing probiotics for 4 weeks. However, measures were not collected in babies during the first month after birth.

In this study we want to test the safety of D-lactate producing bacteria in babies from birth to 1 month of age. This safety study is a randomized, controlled, single center, clinical trial of 2 groups of infants.

The primary objective of this clinical trial is:

to evaluate the effect of a starter formula containing D-lactate producing probiotics versus a starter formula without probiotics, on D-lactic acid urine levels in healthy formula-fed infants, from birth to 28 days of age. Urinary D-lactate concentration (mmol/mol creatinine), will be measured at (baseline, 7 days, 14 days and 28 days).

Secondary objectives include evaluation of effects on gut microbiota, gastrointestinal tolerance, duration of sleep and crying, morbidity and growth, with a follow up to 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies, full term (≥37 weeks gestation) who are 0-24 hours of age at enrolment.
* Babies anticipated to be exclusively formula-fed.
* Babies under the care of a paediatrician or other qualified healthcare professional and have had at least one postnatal visit.
* Study explained and written information provided to Parent/Caregiver demonstrating understanding of the given information.
* Informed consent signed (parent/legal representative)

Exclusion Criteria:

* Babies with chromosomal or major congenital anomalies.
* Significant pre natal and/or post natal disease
* Babies receiving an antibiotic
* Babies born from mothers using supplemental probiotics during the last trimester of pregnancy and/or antibiotics during the last 14 days of pregnancy.
* Babies' family, of whom in the investigator's assessment, cannot be expected to comply with the protocol.
* Babies currently participating in another clinical study

Ages: 1 Hour to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
D-lactic acid urine measure in babies | 1 month

SECONDARY OUTCOMES:
anthropometric measures (Weight, length, and head circumference, stool microbiota, adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Helena Venizelou, Athens, Greece

REFERENCES:
- [Derived] Garcia Rodenas CL, Lepage M, Ngom-Bru C, Fotiou A, Papagaroufalis K, Berger B. Effect of Formula Containing Lactobacillus reuteri DSM 17938 on Fecal Microbiota of Infants Born by Cesarean-Section. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):681-687. doi: 10.1097/MPG.0000000000001198. PMID 27035371